CLINICAL TRIAL: NCT03427229
Title: Randomized Clinical Trial: Single Versus Multiple-infusion Fecal Microbiota Transplantation for Severe Clostridium Difficile Infection
Brief Title: Fecal Microbiota Transplantation for Severe Clostridium Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giovanni Cammarota, Associate Professor of Gastroenterology, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1206132017
Record Dates: First submitted 2017-11-08; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Clostridium Difficile; Pseudomembranous Colitis
Keywords: fecal microbiota transplantation; Clostridium difficile infection; pseudomembranous colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple-infusion FMT (Experimental): Repeated fecal infusions by colonoscopy. Before FMT, vancomycin is administered in all patients for 3 days
  Interventions: Drug: Vancomycin (before randomization); Biological: multiple-infusion FMT
- Single-infusion FMT (Active Comparator): Single fecal infusion by colonoscopy.Before FMT, vancomycin is administered in all patients for 3 days
  Interventions: Biological: Single-infusion FMT; Drug: Vancomycin (before randomization)

INTERVENTIONS:
Biological: Single-infusion FMT — Patients will receive a single fecal infusion by colonoscopy
  Arms: Single-infusion FMT
Drug: Vancomycin (before randomization) — Vancomycin is administered in all patients for 3 days before randomization. Then vancomycin is stopped and patients are randomized to single-infusion FMT or multiple-infusion FMT.
Biological: multiple-infusion FMT — Patients will receive multiple fecal infusions by colonoscopy
  Arms: Multiple-infusion FMT

SUMMARY:
Fecal microbiota transplantation (FMT) is acknowledged as a highly effective treatment for recurrent Clostridium difficile infection (CDI). Usually single fecal infusion achieves satisfactory cure rates of recurrent CDI). However, several retrospective studies show that severe clinical picture of recurrent CDI is a risk factor for the failure of single-infusion FMT, suggesting that multiple fecal infusions are required to cure this condition.

This is an open-label randomized clinical trial aiming to assess if multiple-infusion FMT is more effective than single-infusion FMT in curing severe CDI

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) is acknowledged as a highly effective treatment for recurrent Clostridium difficile infection (CDI). Usually single fecal infusion achieves satisfactory cure rates of recurrent CDI). However, several retrospective studies show that severe clinical picture of recurrent CDI is a risk factor for the failure of single-infusion FMT, suggesting that multiple fecal infusions are required to cure this condition.

This is an open-label randomized clinical trial aiming to assess if multiple-infusion FMT is more effective than single-infusion FMT in curing severe CDI

The investigators' study is an open-label randomized controlled trial, enrolling patients with recurrent and refractory C. difficile infection with a severe clinical picture of the disease.

At enrollment, C. difficile infection is defined as diarrhoea (at least 3 loose or watery stools per day for 2 or more consecutive days, or at least 8 loose stools in 48 hours) and positivity in the C. difficile toxin stool test.

Recurrent C. difficile infection is meant as the reappearance of clinical symptoms and positivity of C. difficile toxin test within 8 weeks after the end of the previous therapy.

Refractory CDI is defined as CDI unresponsive to the antimicrobial treatment, namely persistence of diarrhoea with CD toxin positive or persistent diarrhoea with toxin negative in the absence of other possible causes of diarrhoea (e.g. IBS, IBD, non-CDI antibiotic-associated diarrhea) Severe CDI is defined, according to the latest ESCMID guidelines, as: Episode of CDI with one or more specific clinical (fever, haemodynamic instability, respiratory failure which needs mechanical ventilation, signs and symptoms of peritonitis, signs and symptoms of colonic ileus), laboratory (marked leukocytosis, rise in serum creatinine and lactate, marked decrease of serum albumin), radiological (colon distension, colonic wall thickening) or endoscopic (pseudomembranous colitis), symptoms and signs of severe colitis or complicated course of disease.

Patients' stool are screened for detection of parasites and enteric bacterial pathogens to exclude other infective pathogens. Patients with former colectomy, inflammatory bowel diseases (IBD), irritable bowel syndrome (IBS), viral hepatitis, AIDS or syphilis will be excluded.

Patients are instructed and invited to signal recurrent symptoms and diarrhea after treatment. Monthly clinical and lab checks are performed for a period of 2 months after the treatment.

Treatment procedures:

All patients start therapy with vancomycin for 3 days before of stratification, with random allocation (1 to 1, through statistical software) to one of the two treatment schemes: 1) single-infusion FMT by colonoscopy, with the infusion in the cecum - through the biopsy channel - of 60-120 gr (depending on production) of donated feces, obtained from the donor within 6 hours from transplantation, and manually homogenized in 100/200 ml of physiological solution; colonoscopy will be performed by an expert endoscopist; preparation for colonoscopy (four liters of a solution with saline laxatives) will be provided 2) multiple-infusion FMT (with the same protocol of the other arm, but with repeated fecal infusions).

All patient will be instructed on hygiene rules to be followed at the patient's domicile to avoid re-infections at home. Stool donors will be selected following recommendations from the European FMT Working Group Consensus Conference.

ELIGIBILITY:
Inclusion criteria:

* Recurrent C. difficile infection (identified by positivity of C. difficile toxin in stools) with severe clinical picture (defined by the ESCMID Guidelines published in 2014 - Debast et al, Clin Microbiol Infect 2014)
* Possibility to undergo standard antimicrobial therapy for recurrent C. difficile infection Approval of informed consent
* Possibility to undergo protocol diagnostic and therapeutic procedures
* Stool negativity for parasites
* Stool negativity for Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogenic Escherichia coli and other microorganisms except for C. difficile
* Blood negativity for: Hepatitis A virus-Immunoglobulin M, HBsAg, Anti-Hepatitis C Virus, Anti-Human Immunodeficiency Virus1-2, venereal disease reaction level (VDRL).

Exclusion Criteria:

* Subjects <18 years old
* Prior colectomy
* Negativity of C. difficile toxin in stools
* Mild clinical picture of C. difficile infection
* High risk of post-colonoscopy complications
* Other main gastrointestinal diseases (es. Crohn's disease or ulcerative colitis)
* Stool positivity for parasites
* Stool positivity for Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogenic Escherichia coli and other microorganisms except for C. difficile
* Blood positivity for: Hepatitis A virus-Immunoglobulin M, HBsAg, Anti-Hepatitis C Virus, Anti-Human Immunodeficiency Virus1-2, venereal disease reaction level (VDRL).
* Pregnancy or breastfeeding.
* Inability to follow protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Cure of C. difficile infection | 8 weeks
  Disappearance of C. difficile-associated diarrhea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ianiro G, Masucci L, Quaranta G, Simonelli C, Lopetuso LR, Sanguinetti M, Gasbarrini A, Cammarota G. Randomised clinical trial: faecal microbiota transplantation by colonoscopy plus vancomycin for the treatment of severe refractory Clostridium difficile infection-single versus multiple infusions. Aliment Pharmacol Ther. 2018 Jul;48(2):152-159. doi: 10.1111/apt.14816. Epub 2018 May 30. PMID 29851107